CLINICAL TRIAL: NCT03379064
Title: Exploratory Randomised Controlled Trial of a Culturally Adapted Psychological Intervention for the Management of Irritable Bowel Syndrome (IBS) in a Low-income Country
Brief Title: Culturally Adapted Psychological Intervention for the Management of Irritable Bowel Syndrome (IBS)
Acronym: IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Collaborators: Karachi Medical and Dental College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PILL-IBS-001
Record Dates: First submitted 2017-10-26; First posted 2017-12-20 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome, Low Income Country
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- culturally adapted Cognitive Behavior Therapy (Experimental): We will use The STreSS CBT manual developed by Schroder and his colleagues
  Interventions: Behavioral: Culturally adapted Cognitive Behavior Therapy for IBS
- Treatment As Usual (No Intervention): The Treatment As Usual (TAU) group will receive regular treatment they have been receiving already as prescribed by the physician.

INTERVENTIONS:
Behavioral: Culturally adapted Cognitive Behavior Therapy for IBS — Culturally adapted Cognitive Behavior Therapy for IBS
  Arms: culturally adapted Cognitive Behavior Therapy

SUMMARY:
Irritable bowel syndrome (IBS) is a highly prevalent functional bowel disorder routinely encountered by healthcare providers although it's not life-threatening, this chronic disorder has ability to reduce patients' quality of life and imposes a significant economic burden to the healthcare system.Despite the high prevalence of IBS and its association with disability and adverse effect on health related quality of life we are not aware of any published trial of psychological intervention for IBS from Pakistan. We aim to test the feasibility and acceptability of culturally adapted Cognitive Behaviour Therapy (CBT) for the management of IBS in Karachi, Pakistan compared to treatment as usual.

DETAILED DESCRIPTION:
A systematic review suggested no overall difference in the rates of IBS in East and West . In a population based study from Pakistan. Prevalence of IBS was assessed using Rome II criteria in relation to psychological distress, disability and life events in men and women separately. The prevalence of Rome II IBS was 13.3% which was higher than most population-based studies in Asia using Rome II criteria and similar to reports from Turkey and Malaysia.The findings also suggest equal sex ratio of IBS in urban Pakistan which may be because of the close association between marked distress and IBS in men similar to that found in women in the west.The results indicated that diarrhea-predominant IBS was associated with less disability compared to the constipation-predominant IBS which was associated with marked disability. This might be explained by the explanatory models; constipation is considered harmful as toxins or other harmful substances are retained within the body whereas diarrhea is not considered harmful as any toxins etc are removed from the body. Distress and life events contributed independently to high disability. In psychological treatments there is an assumption that there are some critical features which need to be addressed in the treatment process such as stress and anxiety; it also suggests that stress has a major role in increasing IBS symptoms as well as stress reactivity which results in IBS symptoms. The goal of cognitive-behavioral treatments is to increase awareness regarding the association between stress, thoughts, and IBS symptoms, it is important to identify and modify cognitive appraisals and to change depressive and/or anxiety-based schema. These interventions play a major role in decreasing IBS symptoms severity and associated anxiety and depression when compared to no treatment or standard medical care.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with ROME 111 diagnoses of IBS
* Between the age bracket of 18 to 55 years.
* willing to give written informed consent.

Exclusion Criteria:

* Individuals with atypical symptoms (rectal bleeding, anaemia or unexplained weightloss).
* Diagnosis of inflammatory bowel disease, celiac disease or colon cancer.
* Pregnant or breast feeding.
* History of drug, alcohol, or chemical abuse within 6 months prior to screening.
* Metabolic dysfunction, serious physical examination finding, or clinical laboratory finding giving reasonable suspicion that it might affect the interpretation of the re-sults or render the patient at high risk from treatment complication

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2017-12-30 (Actual); Primary Completion 2018-10-20 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
IBS-symptom severity scale | Change to baseline at 3rd Month
  The score of this system is based on five items (severity and duration of pain, abdominal distension, bowel satisfaction, and interference with life in general) and uses visual analogue scales. Patients can be categorized as having mild (75-175), moderate (175-300), or severe (>300) IBS.

SECONDARY OUTCOMES:
IBS Rome III | Baseline
  IBS symptoms will be recorded using Rome III Modular Questionnaire
IBS quality of Life III | Baseline & 3rd Month
  The IBS-Qol is a 34-item measure of the degree to which IBS symptoms affect lives (5-point scale) The individual responses to the 34 items are summed and averaged for a total score and then transformed to a 0-100 scale for ease of interpretation with higher scores indicating better IBS specific quality of life. There are also eight subscale scores for the IBS-QOL (Dysphoria, Interference with Activity, Body Image, Health Worry, Food Avoidance, Social Reaction, Sexual, Relationships).
IBS pain scale-Pain Vigilance and Awareness Questionnaire | Baseline & 3rd Month
  This 16-item measure will be used to assess pain awareness on a 0-5 point scale, tapping into constructs of awareness, vigilance, preoccupation, and observation of pain. Participants will rate a number of statements from 0 (Never) to 5 (Always) such as; I keep track of my pain level.
Brief Disability Questionnaire (BDQ) | Baseline & 3rd Month
  Disability will be assessed using the cross-culturally validated BDQ, which includes 6 items from the SF-36, asking subjects whether they had been limited in various everyday activities during the last month and four ques-tions concerning daily functioning. Total scores across items 1-6 are considered to indicate 'moderate' and 'severe' disability for score ranges 8-13 and 14-22 respectively. Additionally, participants were asked to estimate how many days over the prior few weeks they were unable to carry out their usual daily activities thus providing an estimate of 'functional disability'.
Client Satisfaction Questionnaire | 3rd month
  CSQ is an 8-item scale that shall be used to measure satisfaction with the treatment received. CSQ is an 8-item scale that shall be used to measure satisfaction with the treatment received.This scale is scored by summing the individual item scores to produce a range of 8 to 32, with high scores indicating greater satisfaction
Global Improvement Scale (GIS) | 3rd month
  Global Improvement will be assessed with the Global Improvement Scale (GIS).This scale asks participants "Compared to the way you felt before you entered the study, have your IBS symptoms over the past 7 days been from (1) = substantially worse, to (7) = substantially improved. Global improvement is noted for patients endorsing moderately or substantially improved status.
EQ-5D (EuroQol-5 Dimensions) | Baseline and 3rd month
  It is a generic measure in which health status is defined in terms of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.Each dimension has three qualifying levels of response roughly corresponding to 'no problems', 'some difficulties/problems', and 'extreme difficulties. The scale has been already used in Pakistan.
Mini International neuropsychiatric Interview (MINI) | Baseline
  Mini International neuropsychiatric Interview (MINI) will be used as a psychiatric diagnostic instrument. It is a short structured diagnostic interview, for DSM-IV and ICD- 10 psychiatric disorders. With an administration time of approximately 15 minutes, it was designed to meet the need for a short but accurate structured psychiatric interview for multicenter clinical trials and epidemiology studies and to be used as a first step in outcome tracking in non research clinical settings.
Hospital Anxiety and Depression Scale (HADS) | Baseline and 3rd month
  The Hospital Anxiety and Depression Scale (HADS) shall be used to assess anxiety and depression. Score 0-7 is considered as (NORMAL) 8 to 10 (Borderline Normal) 11-14 (Moderate), 15 to 21 (Severe) for sub scale separately
The Illness Perception Questionnaire (IPQ) | Baseline
  The IPQ will be used to assess the cognitive representations of illness. The Identity scale is comprised of 12 core symptom items that the patient is asked to rate for frequency on a four point scale ranging from "all of the time" to "never". There are total 26 items in rest of the 4 scales and are rated by the patient on a five point scale ranging from "Strongly Disagree" to "Strongly Agree" (scored 1 to 5)
Short Explanatory Model Interview | Baseline
  SEMI is a short interview that will be administered to elicit the explanatory models.The interview explores the participants' cultural background, nature of presenting problem, help seeking behaviours, interaction with physician and beliefs related to illness.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Nusrat Husain, Principal Investigator — University of Manchester
Locations (1):
- Abasi Shaheed Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No